CLINICAL TRIAL: NCT01165541
Title: An Open-Label, Sequential Study of Quetiapine Fumarate Extended Release (XR) and Mirtazapine for the Treatment of Alcohol Dependency in Very Heavy Drinkers
Brief Title: A Study of Quetiapine and Mirtazapine for the Treatment of Alcohol Dependency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Alan Green, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: QM1
Record Dates: First submitted 2010-07-16; First posted 2010-07-20 (Estimated); Results first posted 2014-03-31 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-03

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — Mirtazapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Quetiapine fumarate extended release (Quetiapine XR) (Active Comparator): Quetiapine XR 50-400mg
  Interventions: Drug: Quetiapine fumarate extended release (Quetiapine XR)
- Quetiapine XR and Mirtazapine (Experimental): Quetiapine XR 50-400mg + Mirtazapine 7.5-45mg
  Interventions: Drug: Mirtazapine; Drug: Quetiapine fumarate extended release (Quetiapine XR)

INTERVENTIONS:
Drug: Mirtazapine — mirtazapine (7.5-45mg)
  Other Names: mirtazapine (Remeron)
  Arms: Quetiapine XR and Mirtazapine
Drug: Quetiapine fumarate extended release (Quetiapine XR) — Quetiapine fumarate extended release 50-400mg/d
  Other Names: quetiapine XR, Seroquel XR

SUMMARY:
The purpose of the study is to test whether taking two medicines (quetiapine and mirtazapine) is better for helping people to decrease drinking than taking one medicine alone (quetiapine).

DETAILED DESCRIPTION:
Alcohol dependence is a debilitating illness affecting almost 8 million people annually and for which the current FDA approved medications are only modestly effective in reducing relapse or drinking. Because alcohol dependence is such a common, devastating disease, researchers continue to search for new treatments that could be more effective and better tolerated. The development and testing of medications that target brain systems involved in alcohol dependence is of acute interest to patients, clinicians and researchers.

Studies by our group in animals have suggested that medications with a combination of a weak dopamine D2 receptor antagonism, a potent norepinephrine alpha 2 receptor antagonism, and norepinephrine reuptake inhibition decrease alcohol drinking. Quetiapine is a weak D2 antagonist and a moderate alpha 2 receptor antagonist, and its primary metabolite, desalkylquetiapine, is a norepinephrine reuptake inhibitor, this medication is likely to have some ability to decrease alcohol drinking. But, when combined with mirtazapine, a potent alpha 2 antagonist, the combination should potently decrease alcohol drinking. The proposed study is based on this theoretical formulation, as well as on clinical studies of quetiapine and mirtazapine used independently.

This is an open-label, sequential design study with one group of approximately 20 subjects studied under two treatment conditions; quetiapine alone and quetiapine + mirtazapine. The primary objective is to assess the efficacy of quetiapine fumarate extended-release (XR) alone vs. quetiapine fumarate XR in combination with mirtazapine in reducing the weekly percentage of days of heavy drinking (5 or more drinks per drinking day for men, 4 or more drinks per drinking day for women) in subjects meeting DSM-IV criteria for alcohol dependency.

Participants will begin with quetiapine fumarate XR up to a target dose of 400 mg and will receive 16 weeks of treatment with quetiapine. At week 8 subjects will begin 9 weeks of mirtazapine added to their existing regimen of quetiapine treatment. Participants will also meet with a medical provider at each visit to encourage compliance with study medication and attending study visits, review adverse events, and set goals for reduction of drinking. Analyses will assess whether treatment with quetiapine in combination with mirtazapine reduces drinking more than treatment with quetiapine alone.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-64
2. The subject meets Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) criteria for alcohol dependence
3. The subject is seeking treatment for alcohol dependence and desires a reduction or cessation of drinking
4. The subject is able to verbalize understanding of the consent form, able to provide written informed consent, and able to verbalize willingness to complete study procedures?
5. If the subject is female and of child bearing potential, she agrees to use an acceptable method of birth control.
6. The subject is able to take oral medication, willing to adhere to the medication regimen, and willing to return for regular visits.
7. The subject is able to understand written and oral instructions in English and able to complete the questionnaires required by the protocol.
8. The subject has a breath alcohol concentration (BAC) equal to 0.000 on s/he signing the informed consent document.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Brunette, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (2):
- United States (2):
  - Dartmouth Medical School Department of Psychiatry's Addition Research Center, Bedford, New Hampshire
  - Dartmouth Medical School Department of Psychiatry's Addiction Research Center, Hanover, New Hampshire

RESULTS

PARTICIPANT FLOW:
Groups:
- Entire Study Population: Quetiapine fumarate extended release (Quetiapine XR): Quetiapine fumarate extended release 50-400mg/d first for 7 weeks; then Quetiapine XR plus mirtazapine: Quetiapine fumarate extended release (50-400mg) plus mirtazapine (7.5-45mg) for 7 weeks.
Period: Quetiapine XR Monotherapy
Arm/Group | Entire Study Population
Started | 20
Completed | 16
Not Completed | 4
Period: Quetiapine XR and Mirtazepine
Arm/Group | Entire Study Population
Started | 16
Completed | 11
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: Entire study population
Groups:
- Entire Study Population: Quetiapine fumarate extended release (Quetiapine XR): Quetiapine fumarate extended release 50-400mg/d first for 7 weeks; then Quetiapine XR and mirtazapine: Quetiapine fumarate extended release (50-400mg) and mirtazapine (7.5-45mg) for 7 weeks.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (10.1)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Very Heavy Drinking Days Per Week
Description: The number of "very heavy" drinking days (8 or more drinks per drinking day for men or 6 or more drinks per drinking day for women) per week
Time Frame: 14 Weeks
Population: The Analysis Population only consists of participants that completed both phases of the study.
Measure: Mean (Standard Deviation); unit: days
Groups:
- Quetiapine XR Plus Mirtazapine: Quetiapine XR 50-400mg + Mirtazapine 7.5-45mg
  Quetiapine XR plus mirtazapine: Quetiapine fumarate extended release (50-400mg) plus mirtazapine (7.5-45mg)
Arm/Group | Quetiapine Fumarate Extended Release (Quetiapine XR) | Quetiapine XR Plus Mirtazapine
Number analyzed (Participants) | 11 | 11
days | 2.1 (2.8) | 1.3 (2.4)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout both periods of the study and included a 30 day follow-up call made after study participation ended to assess for additional events..
Description: This study included two phases (quetiapine XR monotherapy and quetipapine XR andmirtazapine). An adverse event was attributed to a given phase if it began during that phase.
Groups:
- Quetiapine XR andMirtazapine: Quetiapine XR 50-400mg + Mirtazapine 7.5-45mg
  Quetiapine XR and mirtazapine: Quetiapine fumarate extended release (50-400mg) and mirtazapine (7.5-45mg)
Arm/Group | Quetiapine Fumarate Extended Release (Quetiapine XR) | Quetiapine XR andMirtazapine
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/16
Other Adverse Events (participants affected / at risk) | 20/20 | 14/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quetiapine Fumarate Extended Release (Quetiapine XR) (N=20) | Quetiapine XR andMirtazapine (N=16)
Prolonged QTC (Cardiac disorders) | 0 (0) | 1 (1)
Dermatological Condition (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dizzy (Nervous system disorders) | 6 (6) | 1 (1)
Unusual Dream Activity (Psychiatric disorders) | 3 (3) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 7 (7) | 2 (2)
Fatigue (General disorders) | 5 (6) | 3 (4)
Foggy Thinking (General disorders) | 3 (4) | 3 (4)
Gastrointestinal Problems (Gastrointestinal disorders) | 9 (12) | 4 (7)
Headache (Nervous system disorders) | 4 (4) | 3 (4)
Insomnia (Nervous system disorders) | 3 (4) | 2 (3)
Irritated (Psychiatric disorders) | 2 (2) | 1 (1)
Miscellaneous Sleep Disorder (Psychiatric disorders) | 2 (2) | 1 (1)
Muscoloskeletal Disorder (Musculoskeletal and connective tissue disorders) | 3 (4) | 7 (10)
Neurologic Disorder (Nervous system disorders) | 4 (5) | 3 (3)
Nose Bleeds (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Psychiatric Symptoms (Psychiatric disorders) | 2 (4) | 2 (2)
Somnolence (Nervous system disorders) | 8 (9) | 6 (6)
Sweats (General disorders) | 1 (1) | 2 (2)
Increase Triglycerides (Investigations) | 0 (0) | 2 (2)
Upper Respiratory Symptoms (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 0 (0)
Weight Gain (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Blurred Vision (Eye disorders) | 1 (1) | 0 (0)
Decreased Smoking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Libido Descreased (Psychiatric disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Appetite Increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 2 (5) | 1 (1)
Swelling (General disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No